CLINICAL TRIAL: NCT00003061
Title: Evaluating the MBVP Chemotherapy Schedule Followed by Consolidating Radiotherapy in Non-AIDS Related Primary Central Nervous System Lymphoma (NAPCL)
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Primary CNS Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-20962; EORTC-20962
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Cytarabine; Methotrexate; Radiotherapy

INTERVENTIONS:
Drug: cytarabine
Drug: methotrexate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of methotrexate and cytarabine plus radiation therapy in treating patients who have primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of methotrexate and cytarabine chemotherapy in combination with whole-brain radiation therapy for patients with non-AIDS related primary central nervous system lymphoma. II. Assess the response rate and safety of this chemotherapy regimen.

OUTLINE: Patients receive the first course of chemotherapy as soon as possible after diagnosis and staging. Methotrexate (MTX) IV is administered over 40-60 minutes on days 1 and 15. Cytarabine (AraC) is administered intrathecally on days 1 and 15. The second course of chemotherapy begins on day 29 or after bone marrow recovery. Radiation therapy begins no later than 3 weeks after completing chemotherapy. Patients are followed until death.

PROJECTED ACCRUAL: A maximum of 50 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven non-Hodgkin's lymphoma of the central nervous system (CNS) including leptomeninges and the spinal cord No Burkitt's lymphoma or low grade T-cell lymphoma Must have at least 1 measurable lesion No AIDS-related primary central nervous system lymphoma (PCNSL) No disease confined to the eye without other localization in the CNS

PATIENT CHARACTERISTICS: Age: 16 to 60 Performance status: Karnofsky 40-100% Neurological functional status 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No serious impairment of hepatic function Renal: No serious impairment of renal function Creatinine no greater than 1.5 mg/dL OR Creatinine clearance no less than 50 mL/min Cardiovascular: No serious impairment of cardiac function Other: HIV negative No congenital or acquired immunodeficiency syndrome No prior/concurrent systemic lymphoma No prior malignancy except: Adequately treated non-melanoma skin cancer Carcinoma in situ of the cervix uteri Not pregnant No severe uncontrolled infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent treatment with immunosuppressive drug Chemotherapy: No prior chemotherapy Endocrine therapy: Corticosteroid use for less than 3 weeks allowed Radiotherapy: Not specified Surgery: No prior organ transplantation

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 1997-07; Primary Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Poortmans, MD, PhD, Study Chair — Dr. Bernard Verbeeten Instituut
Locations (7):
- U.Z. Gasthuisberg, Leuven, Belgium
- Institut Gustave Roussy, Villejuif, France
- Netherlands (5):
  - Atrium Medical Centre, Heerlen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Rotterdam Cancer Institute, Rotterdam
  - Dr. Bernard Verbeeten Instituut, Tilburg
  - Academisch Ziekenhuis Utrecht, Utrecht

REFERENCES:
- [Result] Harder H, Holtel H, Bromberg JE, Poortmans P, Haaxma-Reiche H, Kluin-Nelemans HC, Menten J, van den Bent MJ. Cognitive status and quality of life after treatment for primary CNS lymphoma. Neurology. 2004 Feb 24;62(4):544-7. doi: 10.1212/wnl.62.4.544. PMID 14981168
- [Result] Poortmans PM, Kluin-Nelemans HC, Haaxma-Reiche H, Van't Veer M, Hansen M, Soubeyran P, Taphoorn M, Thomas J, Van den Bent M, Fickers M, Van Imhoff G, Rozewicz C, Teodorovic I, van Glabbeke M; European Organization for Research and Treatment of Cancer Lymphoma Group. High-dose methotrexate-based chemotherapy followed by consolidating radiotherapy in non-AIDS-related primary central nervous system lymphoma: European Organization for Research and Treatment of Cancer Lymphoma Group Phase II Trial 20962. J Clin Oncol. 2003 Dec 15;21(24):4483-8. doi: 10.1200/JCO.2003.03.108. Epub 2003 Nov 3. PMID 14597741
- [Result] Kluin-Nelemans JC, Poortmans P, Haaxma-Reicher H, et al.: Final results of the EORTC phase II trial 20962 evaluating high-dose MTX-based chemotherapy followed by consolidating radiotherapy in non-Aids related primary central nervous system lymphoma. [Abstract] Blood 100 (11 pt 1): A-3071, 776a, 2002.